CLINICAL TRIAL: NCT06684054
Title: Study of the Features of Senescent T Lymphocytes Induced by Chemotherapy and Its Relationship with the Efficacy of Neoadjuvant Chemotherapy in Young Triple-negative Breast Cancer Patients, a Single-center, Observational Study.
Brief Title: Studying the Senescent T Cell Features and Its Relationship with the Chemotherapy Efficacy in Young TNBC
Acronym: STFREiYTNBC
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-LCYJ-PY-12
Record Dates: First submitted 2024-02-21; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2023-12

CONDITIONS: T-Cell Dysfunction; Chemotherapy Effect; Adverse Events
Keywords: breast cancer; senescence; chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Anthracyclines; Cyclophosphamide; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The collected blood and tissue samples are frozen in the -80℃ refrigerator or liquid nitrogen tank in our hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NAC group: Participants will receive 6 cycles of TEC/TAC neoadjuvant chemotherapy, and radical mastectomy after chemotherapy. Clinicopathological data, chemotherapy-related adverse events and prognostic information of patients should be collected during the study. 5ml peripheral venous blood will be collected before chemotherapy, after 2 cycles of chemotherapy, before surgery, and six months after surgery.
  Interventions: Drug: docetaxel, anthracycline, cyclophosphamide

INTERVENTIONS:
Drug: docetaxel, anthracycline, cyclophosphamide — 1. Participants were required to receive 6 cycles of TEC/TAC neoadjuvant chemotherapy, and radical mastectomy was required after chemotherapy.
  2. 5ml peripheral venous blood was collected before chemotherapy, after 2 cycles of chemotherapy, before surgery, and six months after surgery.
  3. Clinicopathological data, chemotherapy-related adverse events and prognostic information of patients should be collected during the study.
  Other Names: G-CSF

SUMMARY:
The goal of this observational study is to learn about the features of senescent T lymphocytes induced by chemotherapy and its relationship with the efficacy of neoadjuvant chemotherapy in young triple-negative breast cancer (TNBC) patients.

The main questions it aims to answer are:

* What are the senescent features of peripheral T lymphocytes in young TNBC patients receiving neoadjuvant chemotherapy and the relationship with the efficacy of neoadjuvant chemotherapy?
* What is the relationship between senescent T cells and adverse events, DFS and tumor infiltrating lymphocytes?

  1. Participants will receive 6 cycles of docetaxel + adriamycin/epirubicin + cyclophosphamide (TEC/TAC) neoadjuvant chemotherapy, and radical mastectomy after chemotherapy.

2.5ml peripheral venous blood will be collected before chemotherapy, after 2 cycles of chemotherapy, before surgery, and six months after surgery.

3.Clinicopathological data, chemotherapy-related adverse events and prognostic information of patients should be collected during the study.

DETAILED DESCRIPTION:
This is a single-center observational study that is expected to enroll 30 breast cancer patients and 10 controls from July 2023 to June 2026. We mainly want to investigated senescent T lymphocytes characteristics during neoadjuvant chemotherapy in young triple-negative breast cancer patients. Besides, the relationship between senescent T lymphocytes and neoadjuvant chemotherapy efficacy also of concern to us.

Inclusion criteria: (1) female, age ≤40 years old; (2) Invasive breast cancer was confirmed by puncture pathology and TNBC (ER-, PR-, HER2-) was confirmed by immunohistochemistry; (3) Patients who meet the indications of neoadjuvant chemotherapy prescribed in the guidelines.

Exclusion criteria: (1) IV patient or history of other malignant tumors; (2) Recently infection or autoimmune disease is not cured or HBV, HIV positive; (3) Had a history of surgery 3 months before enrollment; (4) Patients with insufficient clinicopathological data; (5) Those who do not meet the evidence of neoadjuvant chemotherapy or are unwilling to cooperate.

Withdrawal criteria: (1) the subjects did not receive radical surgery in our hospital or were unwilling to continue to participate in the follow-up study; (2) Termination of chemotherapy due to serious side effects or disease progression during chemotherapy; (3) Research data related to the experiment is missing and cannot be supplemented; (4) Poor specimen quality (hemolysis, contamination, etc.); (5) Follow-up lost.

Participants will receive 6 cycles of TEC/TAC neoadjuvant chemotherapy, and radical mastectomy after chemotherapy. Clinicopathological data, chemotherapy-related adverse events and prognostic information of patients should be collected during the study. 5ml peripheral venous blood will be collected before chemotherapy, after 2 cycles of chemotherapy, before surgery, and six months after surgery. The senescence phenotype of T lymphocytes will be determined by flow cytometry.

The main purpose are:

* Studying the senescent features of peripheral T lymphocytes in young TNBC patients receiving neoadjuvant chemotherapy and the relationship with the efficacy of neoadjuvant chemotherapy.
* Studying the relationship between senescent T cells and adverse events, DFS and tumor infiltrating lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age≤40 years old,
2. Invasive breast cancer confirmed by pathology, immunohistochemistry showed TNBC (ER-, PR-, HER2-),
3. Indications for neoadjuvant chemotherapy according to guidelines: tumor diameter > 2cm or with axillary lymph node metastasis or desiring breast-conserving surgery but should obtain negative surgical margins through neoadjuvant chemotherapy.

Exclusion Criteria:

1. Stage IV patients or a history of other malignancies,
2. Having microbial infection or autoimmune disease have not been cured or having HBV, HIV infection,
3. Having surgery 3 months before enrollment,
4. Patients with insufficient clinicopathological data,
5. Does not meet the indications for neoadjuvant chemotherapy or is unwilling to cooperate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young triple negative breast cancer patients receiving neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR | 2024/7-2027/6
  pathological complete response

IPD SHARING:
Plan to Share IPD: No